CLINICAL TRIAL: NCT07214636
Title: Development and Investigation of the Effectiveness of a Digital Video-Based Game Exercise System (ApneaTheraPlay) for Individuals With Obstructive Sleep Apnea Syndrome
Brief Title: Development and Investigation of the ApneaTheraPlay
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Gülay Aras Bayram, PhD, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-10840098-202.3.02-6266
Record Dates: First submitted 2025-09-23; First posted 2025-10-09 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Apnea, Obstructive; Exercise Addiction; Physiotherapy and Rehabilitation
Keywords: Apnea; Exercise; Exergame; Physiotherapy and Rehabilitation; CPAP
MeSH Terms: conditions — Sleep Apnea, Obstructive; Apnea; Motor Activity

STUDY DESIGN:
Intervention Model Description: The randomized controlled, single-blind study
Who Masked: Outcomes Assessor
Masking Description: The researchers performing the assessments and the statistician performing the statistical analysis will be blinded to the group assignments.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Structured Pre-Sleep Exercise Group (SPEG) (Experimental): Individuals will complete a program consisting of 5-minute breathing, 10-minute aerobic, 5-minute strengthening, and 10-minute oropharyngeal exercises, three times a week for 12 weeks, for a total of 36 sessions.
  Interventions: Behavioral: Structured Pre-Sleep Exercise
- ApneaTheraPlay (ATP) Group (Experimental): Participants will exercise individually at pre-sleep times, three days a week, for 12 weeks, using a digital video-based game exercise system developed by researchers, for a total of 36 sessions.
  Interventions: Behavioral: ApneaTheraPlay (ATP)
- Control Group (CG) (No Intervention): Participants in this group will use a physician-prescribed Continuous Positive Airway Pressure (CPAP) device and sleep with CPAP every night for 12 weeks. After the study is completed, participants in this group will also be turned on to the ApneaTheraPlay system and will be encouraged to practice the exercises.

INTERVENTIONS:
Behavioral: Structured Pre-Sleep Exercise — Participants in this group will undergo a new program structured around exercises typically used individually or in combination in the literature, at pre-sleep times. Individuals will complete a program consisting of 5-minute breathing, 10-minute aerobic, 5-minute strengthening, and 10-minute oropharyngeal exercises, three times a week for 12 weeks, for a total of 36 sessions. Two-minute rest breaks will be provided between exercises. The exercises will be presented to users weekly as a video/training sheet prepared by the therapist. Individuals in this group will be monitored and tracked through the system to be developed. This group will only have access to this video/training sheet information in the user panel opened in the system. The system will remind users of the exercises as an exercise program, without gamification, and will provide instant data flow.
  Arms: Structured Pre-Sleep Exercise Group (SPEG)
Behavioral: ApneaTheraPlay (ATP) — Participants will exercise individually at pre-sleep times, three days a week, for 12 weeks, using a digital video-based game exercise system developed by researchers, for a total of 36 sessions. Access to the exercise program will be provided via a web system, and all time spent in the system and reactions will be recorded in a report. The ApneaTheraPlay system will implement programs consisting of breathing (5 minutes), aerobic (10 minutes), strengthening (5 minutes), and oropharyngeal exercises (10 minutes) in a predetermined progression.
  Arms: ApneaTheraPlay (ATP) Group

SUMMARY:
Obstructive Sleep Apnea Syndrome (OSAS) is commonly treated with CPAP devices, but adherence rates are low. Exercise has been shown to strengthen respiratory muscles, improve upper airway function, and enhance sleep quality. However, most studies have examined only single or dual exercise protocols, and there is little evidence regarding integrated programs with four exercise types or their effects when performed directly before sleep.

This project aims to develop and evaluate ApneaTheraPlay (ATP), a digital gamified video-based exercise platform combining respiratory, aerobic, strengthening, and oropharyngeal exercises. The randomized controlled, double-blind study will allocate participants into three groups: ATP, a structured pre-sleep exercise group (SPEG), and a control group (CG). Intervention groups will exercise three times per week for 12 weeks, while the control group will only keep a physical activity diary.

DETAILED DESCRIPTION:
Obstructive sleep apnea syndrome (OUAS) is a common sleep disorder caused by recurrent collapse of the upper airways during sleep. Continuous positive airway pressure (CPAP) devices are one of the most widely used clinical modalities for treatment. However, the literature reports that compliance with CPAP is low, with non-compliance rates ranging from 46% to 83%. As an alternative and supportive method, exercise has been proven to have positive effects on strengthening respiratory muscles, improving upper airway function and improving sleep quality. Recent studies generally focus on single or dual combined exercise protocols, but there is no comprehensive study on the integrated application of four different exercise types. Furthermore, there is limited evidence in the literature on the efficacy of performing exercises directly before sleep.

This project aims to develop and evaluate the effectiveness of a digital video-based gaming exercise platform (ApneaTheraPlay) that combines respiratory, aerobic, strengthening, and oropharyngeal exercises for individuals with OUAS. The project is designed to increase individual participation in the exercises and maintain patient motivation by using a web-based system that can be applied in the home environment prior to sleep.

The outcome of this project will be the development of a digital, video-based, gamified exercise application for people with OUAS that will both increase exercise compliance and support the effectiveness of CPAP use. In addition, the developed system will enable remote patient monitoring and guidance by providing a virtual clinical environment. This innovative approach to the literature will make an important contribution to the scientific evaluation of the effect of pre-sleep exercise on OUAS symptoms.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age
* Individuals diagnosed with mild, moderate, or severe OSAS (AHI 5-30 events/hour) based on laboratory diagnostic polysomnography assessments
* Individuals diagnosed by a pulmonologist within the last year and who have started CPAP therapy for at most 12 months and who are regular users
* Those with habitual snoring
* All participants in the exercise group must have or have access to a phone, tablet, or computer compatible with SMART technologies using the exercise system app
* Participants must have sufficient physical function to follow the exercise instructions
* Familiarity with mobile health applications, as assessed by the VAS, and a willingness to participate in these exercises of >7
* Not having participated in physiotherapy-based interventions targeting OSAS in the last 3 months
* A score of 68 or higher on the System Usability Scale (SUS)

Exclusion Criteria:

* • BMI > 40 kg/m2

  * Serious drug or alcohol abuse
  * Regular use of sedatives, muscle relaxants, or opioids that may affect sleep patterns or exercise performance
  * Pregnancy or postpartum (<6 months) due to hormonal effects on sleep and respiratory function
  * Any medical contraindication to physical activity (unstable coronary disease, decompensated heart failure) according to the American College of Sports Medicine (ACSM) exercise guidelines (American College of Sports Medicine, 2021)
  * History of stroke
  * Presence of any significant respiratory, neuromuscular, or other disorder causing hypercapnia
  * Systemic disease associated with an inflammatory entity (e.g., arthritis, sarcoidosis, vasculitis, lupus)
  * Craniofacial deformity
  * Presence of secondary respiratory diseases such as severe upper airway obstruction or COPD
  * Presence of dysphagia
  * Presence of a frenulum restricting tongue movement

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2026-05-02 (Estimated); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Apnea-hypopnea index (AHI) | 0.,12., and 24. weeks
  This will be measured objectively during a Level 1 sleep study (polysomnography). The AHI measures the number of apnea and hypopnea events per hour of sleep; 0 to 4 events indicates normal, 5 to 14 events indicates mild OSAS, 15 to 30 events indicates moderate OSAS, and greater than 30 events indicates severe OSAS. A change in AHI of at least 15 events will be considered clinically significant to determine the clinical effectiveness of the intervention.

SECONDARY OUTCOMES:
Oxygen saturation (SaO₂) | 0.,12., and 24. weeks
  This is the percentage of hemoglobin in the blood that is saturated with oxygen. It is a key indicator of respiratory function. As part of the project, participants will be provided with a Huawei GT3 Pro smartwatch (Huawei Technologies Co., Ltd., Shenzhen, China). The smartwatch will monitor and record individuals' SaO₂ levels day and night. A normal oxygen saturation level generally ranges from 95% to 100%, while values below 90% indicate hypoxia. Data from the watch will be used for comparison and follow-up with data from polysomnography.
Pittsburgh Sleep Quality Index (PSQI) | 0.,12., and 24. weeks
  The PSQI is a widely recognized 19-item self-report questionnaire used to assess subjective sleep quality and disturbances over a month. Subjective sleep quality assesses multiple dimensions of sleep, including sleep latency, duration, efficiency, disturbances, use of sleeping pills, and daytime dysfunction. Each component is scored on a scale of 0 to 3, and the total score ranges from 0 to 21; higher scores indicate poorer sleep quality. Scores above 5 are indicative of poor sleep quality.
The Insomnia Severity Index (ISI) | 0.,12., and 24. weeks
  This is a widely used self-report questionnaire designed to assess the severity of insomnia symptoms and their impact on daily functioning. It consists of seven items, each rated on a five-point Likert scale (0-4), and assesses difficulties falling asleep, staying asleep, early morning awakening, sleep dissatisfaction, interference with daytime activities, perception of sleep problems by others, and distress caused by sleep difficulties. The total ISI score ranges from 0 to 28, with higher scores indicating more severe insomnia symptoms. Scores are categorized as follows: no clinically significant insomnia (score of 0-7); subthreshold insomnia (score of 8-14); moderate insomnia (score of 15-21); and severe insomnia (score of 22-28).
Epworth Sleepiness Scale (ESS) | 0.,12., and 24. weeks
  This is a self-report questionnaire designed to assess daytime sleepiness. The ESS consists of eight items, each rated on a 4-point scale (0-3), and measures the likelihood of falling asleep during activities such as reading, watching television, sitting in a public place, or traveling as a passenger. The total score ranges from 0 to 24, with higher scores indicating greater levels of daytime sleepiness. A score of 0-10 is considered normal, while scores above 10 indicate varying degrees of excessive daytime sleepiness.
Functional Sleep Outcomes Questionnaire (FOSQ-10) | 0.,12., and 24. weeks
  A 10-item self-reported questionnaire designed to assess the impact of sleepiness on alertness, activity level, general productivity, social outcomes, and intimate and sexual relationships. Items are rated on a 4-point scale (no difficulty, little difficulty, moderate difficulty, and severe difficulty). A mean score is calculated for each subscale, and the five subscales are summed to yield a total score ranging from 5 to 20, with higher scores indicating better functional status.
Subjective sleepiness and sleep quality | 0.,12., and 24. weeks
  A Visual Analog Scale (VAS) ranging from 0 (not at all sleepy, fully awake and alert) to 10 (excessively sleepy, about to fall asleep) will be assessed three times a day (9:00 AM, 12:00 PM, and 8:00 PM) throughout the study, integrated into the web-based application. Participants' subjective sleep quality will be assessed daily upon awakening using a Visual Analog Scale (VAS) ranging from 0 to 10, integrated into the developed web-based system. On this scale, 0 represents "very poor" and 10 represents "very good" sleep quality.
The Chalder Fatigue Scale (CFS) | 0.,12., and 24. weeks
  This 11-item scale was developed to measure the severity of fatigue in adults. It is used in both clinical and research settings. Fatigue-related items are scored on one of four Likert-type responses: "better than usual," "not better than usual," "worse than usual," or "much worse than usual."
MIP-MEP measurement | 0.,12., and 24. weeks
  In centimeters of water (cmH2O), it will be obtained using a Respiratory Muscle Strength Measurement Device-MIP-MEP (MD Diagnostics Ltd., RP Check, United Kingdom) in accordance with the recommendations of the American Thoracic Society.
Forced Vital Capacity (FVC) measurement | 0.,12., and 24. weeks
  It is the amount of air expelled after maximum inspiration following a normal breath, expressed in liters. While healthy individuals can forcefully exhale air for 2-3 seconds, this time can be as short as 10-15 seconds for individuals with airway problems. At the end of the test, the expected reference value should be between 80-120%.
  This will be performed using a spirometer (Cosmed, Pony FX, Italy). The best forced vital capacity (FVC) maneuver from at least 3 attempts will be selected according to the criteria of the American Thoracic Society. To perform the spirometric maneuvers, participants will sit upright with their feet on the floor and the nose clip correctly positioned.
FEV₁ (Forced Expiratory Volume in 1 Second) | 0.,12., and 24. weeks
  It is the volume of air exhaled in the first second after forced expiration. Although measured in liters, it actually indicates the airflow rate. In healthy individuals, at least 72% of the air should be exhaled, reflecting the function of the large airways.
  This will be performed using a spirometer (Cosmed, Pony FX, Italy). To perform the spirometric maneuvers, participants will sit upright with their feet on the floor and the nose clip correctly positioned.
FEV1/FVC ratio | 0.,12., and 24. weeks
  This ratio is obtained by dividing FEV1 by FVC and evaluates airway patency and lung function. In a normal individual, this ratio is around 70-80%.
  This will be performed using a spirometer (Cosmed, Pony FX, Italy). To perform the spirometric maneuvers, participants will sit upright with their feet on the floor and the nose clip correctly positioned.
FEF 25%-75% (Maximal Mid-Expiratory Flow Rate) | 0.,12., and 24. weeks
  It refers to the average airflow rate during forced expiration, when 25% to 75% of the volume is expelled. It is measured in liters per second. It reflects the function of the medium and small airways. A value above 80% of the reference value is normal.
  This will be performed using a spirometer (Cosmed, Pony FX, Italy). To perform the spirometric maneuvers, participants will sit upright with their feet on the floor and the nose clip correctly positioned.
CPAP adherence data | 0-24. weeks
  The average nightly CPAP usage time from CPAP devices will be recorded. Good CPAP adherence is generally defined as ≥ 4 hours/night for ≥ 5 nights per week.
Exercise Compliance | 0-24. weeks
  The total time participants spend logging into the ApneaTheraPlay system and playing the games will be recorded.
Daily step count | 0-24. weeks
  The weekly step count average will be recorded. Data recorded on the Huawei GT3 Pro smartwatch (Huawei Technologies Co., Ltd., Shenzhen, China) will be collected from users and used for analysis.
Day and night SaO₂ levels | 0-24. weeks
  The minimum and maximum SAO2 values during the day and night will be recorded. Data recorded on the Huawei GT3 Pro smartwatch (Huawei Technologies Co., Ltd., Shenzhen, China) will be collected from users and used for analysis.
Heart rate variability (HRV) | 0-24. weeks
  Heart rate changes during games and exercises will be recorded, from the smallest to the largest values. Data recorded on the Huawei GT3 Pro smartwatch (Huawei Technologies Co., Ltd., Shenzhen, China) will be collected from users and used for analysis.
System Usability Scale (SUS) | 0.week
  It consists of 10 statements that allow you to assess the ease of use (or lack thereof) of websites, software, hardware, mobile devices, and other technological applications at a glance. The SUS is essentially a survey designed to assess usability, using a 5-point Likert scale. The following formula will be used to calculate the SUS score:
  Statements are scaled from 0 to 4 (strongly disagree = 0, strongly agree = 4). First, the score assigned to odd-numbered statements is subtracted from 1 (X-1).
  The score assigned to even-numbered statements is subtracted from 5 (5-X). The calculated items are summed and multiplied by 2.5. The average SUS score is taken as 68, and a SUS score greater than 68 indicates that the system is above average, while a score below 68 indicates that the system is below average. Products with the highest usability ratings are classified as A+, with a percentile range between 96 and 100.
Short Form-12 (SF-12) | 0.,12., and 24. weeks
  In the study, SF-12 Health Survey will be used to assess the general health status and quality of life of individuals. The survey consists of 12 items that assess health status in terms of physical and mental health components. Similar to SF-36, SF-12 also consists of a total of 12 items in 8 subscales: physical functioning, role-physical, bodily pain, general health, energy, social functioning, role-emotional, and spiritual health. The items in the role-physical and role-emotional items are dichotomous and can be answered with "yes" or "no", while the other items are Likert-type with response options between 3 and 6. The scores range from 0 to 100, with higher scores indicating better health status. Higher scores on the SF-12 Health Survey indicate a better quality of life.
Quadriceps isometric muscle strength | 0.,12., and 24. weeks
  Isometric muscle strength for unilateral knee extension will be measured using a myometer (Pelican products, Torrance, CA USA). Participants will be seated in a chair with their hips and knees flexed to 90°, and their hands will be crossed at their sides or across their chest to maintain a stable position. The myometer will be placed on the distal anterior surface of the tibia, a few cm above the malleolus, and the device will be held steady by a physical therapist. Participants will be instructed to "Push your knee forward and up as hard as you can and hold this position for 3-5 seconds." Three repetitions will be performed, with the highest value recorded as quadriceps muscle strength. Measurements will be recorded in kilograms of force (kgf) and will be evaluated separately for both the right and left sides.
Hand Grip Strength | 0.,12., and 24. weeks
  Maximum grip strength will be measured on the dominant arm using a hand dynamometer (Jamar Hydraulic Hand Dynamometer, Sammons Preston CO, Bolingbrook, IL, USA). Participants will be instructed to squeeze the dynamometer as hard as possible while sitting upright, arms at their sides, elbows flexed to 90°, and forearms in a neutral position. Maximum strength will be measured three times with a 2-minute rest between assessments, with the highest value considered the maximum strength.
The Hospital Anxiety and Depression Scale (HADS) | 0.,12., and 24. weeks
  This scale contains a total of 14 questions, with seven odd-numbered questions measuring anxiety and seven even-numbered questions measuring depression. The scale is a four-point Likert-type assessment tool, with item scores ranging from 0 to 3. The lowest possible score for either subscale is 0, and the highest is 21. Studies conducted in Türkiye have found a cutoff score of 10 for the anxiety subscale and 7 for the depression subscale. Individuals scoring above these scores can be considered at-risk.

CONTACTS AND LOCATIONS:
Overall Officials: Gülay Aras Bayram, Principal Investigator — Medipol University
Locations (1):
- Istanbul Medipol Universty, Istanbul, Göztepe Neighborhood, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No